CLINICAL TRIAL: NCT02777814
Title: An Open, Randomized Controlled Clinical Trial to Compare the Prophylactic Use or Preemptive Use of an Anti-viral Drug Entecavir in Patients With Colorectal Cancer Who Are Inactive Hepatitis B Carriers
Brief Title: Prophylactic or Preemptive Entecavir in Patients With Colorectal Cancer Who Are Inactive Hepatitis B Carriers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRC-HBV
Record Dates: First submitted 2016-04-01; First posted 2016-05-19 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; Entecavir; Hepatitis B Carrier
MeSH Terms: conditions — Colorectal Neoplasms | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic Entecavir (Experimental): Entecavir is prophylactically used from the time of chemotherapy initiation at the dose of 0.5 mg p.o daily
  Interventions: Drug: Entecavir
- Preemptive Entecavir (Active Comparator): Entecavir is preemptively used from the time that hepatitis B virus DNA copies are more than 100 IU/ml at the dose of 0.5 mg p.o daily
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — anti hepatitis B virus
  Other Names: Entecavir Dispersible Tablets

SUMMARY:
There has been no report on whether the patients with colorectal cancer who are also inactive Hepatitis B Carriers should receive Prophylactic Use or preemptive Use of an Anti-viral Drug Entecavir. This open, randomized controlled clinical trial aims to compare the impact of the prophylactic use or preemptive use of an anti-viral drug Entecavir on the outcomes of patients with colorectal cancer who are also inactive hepatitis B carriers during chemotherapy and the subsequent follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 18 and 75
2. Patient with histology-proven colorectal adenocarcinoma.
3. Patients with Eastern Cooperative Oncology Group performance status (ECOG) of 0-1
4. Patients planned for at least 4 cycles of cytotoxic chemotherapy (either as part of curative therapy or as palliative therapy)
5. Patients with at least 6 months' life expectancy from date of recruitment
6. Patients with positive Hepatitis B Surface-antigen (HBsAg)
7. Patients with normal liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase alkaline (AST), phosphatase (ALP), gamma glutamyl-transpeptidase (GGT), and bilirubin
8. Patients with negative HBV-DNA
9. Patients with no known history of radiological &/or histological diagnosis of chronic active hepatitis or cirrhosis of any cause, or history of prior hepatitis B reactivation, or prior chronic therapy for HBV within 6 months
10. Patients with no evidence of autoimmune hepatitis, hepatitis C or D virus infection, HIV infection or radiological evidence of liver metastasis
11. adequate bone marrow, hepatic, and renal function within 14 days before recruitment
12. patients who sign the informed consent
13. Patients with good compliance during chemotherapy and follow-ups

Exclusion Criteria:

1. Patients planned for radiation or radionuclide therapy
2. Pregnant female patients
3. Patients with a history of psychiatric drugs abuse and can't quit or with a mental disorder
4. Patients with immunodeficiency, other congenital or acquired immunodeficiency, or transplantation history
5. According to the investigators' judgment, patients with concomitant disease that seriously harms patients' safety or the completion of study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatitis B virus associated hepatitis | through study completion, an average of 1 year
  Hepatitis is defined as a 3-fold or greater increase in the serum ALT level that exceeded the reference range (>58U/L) or an absolute increase in the level of ALT of greater than 100 U/L compared with the baseline level

SECONDARY OUTCOMES:
Incidence of hepatitis B virus reactivation | through study completion, an average of 1 year
  Reactivation of HBV is defined as a 10-fold or greater increase in the HBV DNA level or an absolute increase of 10^5 copies/mL or greater compared with the baseline value.
Interruption of chemotherapy due to hepatitis | through study completion, an average of 1 year
  Chemotherapy disruption is defined as either premature termination or a delay of at least 7 days between chemotherapy cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, M.D. Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Di Bisceglie AM, Lok AS, Martin P, Terrault N, Perrillo RP, Hoofnagle JH. Recent US Food and Drug Administration warnings on hepatitis B reactivation with immune-suppressing and anticancer drugs: just the tip of the iceberg? Hepatology. 2015 Feb;61(2):703-11. doi: 10.1002/hep.27609. PMID 25412906
- [Result] Huang H, Li X, Zhu J, Ye S, Zhang H, Wang W, Wu X, Peng J, Xu B, Lin Y, Cao Y, Li H, Lin S, Liu Q, Lin T. Entecavir vs lamivudine for prevention of hepatitis B virus reactivation among patients with untreated diffuse large B-cell lymphoma receiving R-CHOP chemotherapy: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2521-30. doi: 10.1001/jama.2014.15704. PMID 25514302
- [Result] Perrillo RP, Gish R, Falck-Ytter YT. American Gastroenterological Association Institute technical review on prevention and treatment of hepatitis B virus reactivation during immunosuppressive drug therapy. Gastroenterology. 2015 Jan;148(1):221-244.e3. doi: 10.1053/j.gastro.2014.10.038. Epub 2014 Oct 31. No abstract available. PMID 25447852